CLINICAL TRIAL: NCT01736839
Title: Ultrasensitive Detection of Reductions in Cystic Fibrosis Airway Inflammation While Using Aztreonam Lysine for Inhalation Solution
Brief Title: Detection of Reductions in Cystic Fibrosis Airway Inflammation While Using Aztreonam Lysine Solution
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: IN-US-205-0171
Record Dates: First submitted 2012-11-15; First posted 2012-11-29 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis in Adults, Chronic Colonization With Pseudomonas Aeruginosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CF adults colonized with Pseudomonas aeruginosa

SUMMARY:
In cystic fibrosis, there is a critical need for better predictors of treatment response. The investigators have identified a panel of white blood cell biomarkers which can be directly measured as a blood test in subjects with cystic fibrosis. These biomarkers predict reduction of airway inflammation and infection more accurately than lung function testing, in patients receiving intravenous antibiotic therapy. In the current study, we hypothesize that this panel of gene biomarkers which can be readily measured from peripheral blood will sensitively predict changes in inflammation when patients receive inhaled antibiotic therapy, specifically Cayston (or inhaled aztreonam lysine). Patients enrolled in the study will have blood drawn before and after a month of inhaled Cayston, in order to test whether genes predict response to Cayston therapy more robustly than do standard measures such as lung function tests.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of cystic fibrosis
* Age 18 years old or greater
* FEV1 percent predicted greater than 25%
* Ability to perform reproducible pulmonary function tests and produce sputum spontaneously
* Chronic bacterial colonization with Pseudomonas aeruginosa with 2 positive cultures in previous 2 years.
* Chronically stable pulmonary condition without evidence of acute pulmonary exacerbation within 14 days prior to screening
* Starting Cayston cycle as part of clinical care.

Exclusion Criteria:

* Presence of a condition or abnormality that, in the opinion of the Principal Investigator (PI), would compromise the safety of the patient or the quality of the data.
* Aztreonam allergy, bronchospasm or other contraindication to use of aztreonam.
* Signs and symptoms of acute pulmonary exacerbation at the time of enrollment or during study.
* Active infection and treatment for non-tuberculous mycobacteria.
* Concomitant use of systemic steroids.
* Use of inhaled antimicrobial agents with activity against Pseudomonas aeruginosa within 28 days prior to Visit 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled subjects will include adults with cystic fibrosis, over the age of 18 years, who are at baseline health and colonized with Pseudomonas aeruginosa, and who are newly prescribed Cayston (aztreonam lysine) for inhalation, or who are resuming use of this drug after 28 days off of inhaled antimicrobial agents with activity against Pseudomonas aeruginosa.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-11; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Gene biomarker panel | 1 month
  Measurement of gene biomarkers by polymerase chain reaction before and after 1 month of Cayston therapy

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | 1 month
  Change in pulmonary function (FEV1) after one month of Cayston therapy
Sputum Bacterial Density | 1 month
  Change in sputum bacterial density after one month of Cayston
C-reactive protein | 1 month
  Change in C-reactive protein after one month of Cayston
Interleukin 8 | 1 month
  Change in serum and sputum interleukin 8 concentrations after one month of Cayston
Patient reported symptom scores | 1 month
  Change in patient reported symptoms after one month of Cayston

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Caceres SM, Sanders LA, Rysavy NM, Poch KR, Jones CR, Pickard K, Fingerlin TE, Marcus RA, Malcolm KC, Taylor-Cousar JL, Nichols DP, Nick JA, Strand M, Saavedra MT. Blood mRNA biomarkers distinguish variable systemic and sputum inflammation at treatment initiation of inhaled antibiotics in cystic fibrosis: A prospective non-randomized trial. PLoS One. 2022 May 5;17(5):e0267592. doi: 10.1371/journal.pone.0267592. eCollection 2022. PMID 35511761